CLINICAL TRIAL: NCT05915845
Title: Effects of Laura Mitchell's Relaxation Versus Papworth Exercise on Dyspnea, Fatigue, and Sleep Quality in Ashmatic Patient
Brief Title: Laura Mitchell's Relaxation Versus Papworth Exercise in Ashmatic Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0314
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Asthmatic
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laura Mitchell's Relaxation technique (Experimental)
  Interventions: Other: Laura Mitchell's Relaxation technique
- Papworth exercise (Active Comparator)
  Interventions: Other: Papworth exercise

INTERVENTIONS:
Other: Laura Mitchell's Relaxation technique — This technique was used to eliminate muscular tension. Patients were taught to contract muscles opposite to the strained muscle groups, eventually to 'cease' shrunken them, and then to roster the position adaptation of the body structure. Patient was comfortably positioned.
  Arms: Laura Mitchell's Relaxation technique
Other: Papworth exercise — The Papworth Method integrates five components, the principal one being specific breathing training:
  • Breathing training, including teaching of appropriate minute and tidal volume and the development of a pattern of breathing suitable to current metabolic activity.
  Elimination of dysfunctional breathing, including hyperinflation and hyperventilation patterns is discussed. A specific Papworth method diaphragmatic breathing technique is taught to replace the use of inappropriate accessory muscles of respiration. When relaxed, is placed on calm slow nasal expiration. Patients are encouraged to "nose-breathe" rather than "mouth-breathe" and eradication or reduction of habits such as yawning, sighing, etc. is taught and practiced.
  Arms: Papworth exercise

SUMMARY:
Asthma is a lung disease that is characterized by airway obstruction that is reversible either spontaneously or with treatment, airway inflammation, and increase airway responsiveness to a variety of stimuli. A wide variety of pharmacological interventions are available nowadays. Apart from that, different Physical therapy techniques increase cardiorespiratory fitness and inspiratory pressure and limit symptoms and restrict medication use. Physical therapy techniques that can be beneficial for an asthmatic patient include Breathing exercises (BE), Inspiratory muscle training (IMT), physical therapy training (PhT), and airway clearance (AC). Laura Mitchell's Relaxation technique and Papworth exercise are advised as an effective nonpharmacological intervention leading to the improvement of symptoms in asthmatic patients. In this study the effects of Laura Mitchell's relaxation technique and Papworth exercise on dyspnea, fatigue, and sleep quality in asthmatic patients will be compared. A randomized clinical trial will be conducted at Laeeque Rafiq Hospital, Lar. Convenient sampling technique will be applied on-patients according to the inclusion criteria. Patients will be allocated through simple random sampling into group A & group B. Group A will be treated with Laura Mitchell's Relaxation technique and Group B will be treated with Papworth exercise. Treatment evaluation will be done after 2 weeks of intervention through Pulse Oximeter, Asthma fatigue scale, Dyspnea 12 scale and Pittsburgh sleep quality index. Data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age group of 20-45 years
* Both male and females
* patients diagnosed with asthma according to GINA guidelines, who had not smoked for at least one year

Exclusion Criteria:

* Patients with the history of acute asthmatic attack in last one month.
* Hemodynamically unstable.
* Cough and active hemoptysis

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Pulse Oximeter | 6 weeks
  Pulse oximetry, measuring SpO2 as a proxy for SaO2 using a non-invasive and simple device, is frequently used to detect low blood oxygen levels. Pulse oximetry has been widely used in non-clinical settings, to detect hypoxemia and inform decisions to escalate care
COPD and Asthma fatigue scale | 6 weeks
  The 21-item COPD and Asthma fatigue scale incorporated items on fatigue associated with respiratory disease and breathing problems. The response options were 1 = never to 5 = very often. COPD and Asthma fatigue scale raw scores were linearly transformed to a 0-100 total scale score, with higher scores indicating greater fatigue
Dyspnea 12 scale | 6 weeks
  D-12 consists of 12 descriptor items on a scale of none (0), mild (1), moderate (2), or severe (3). It provides an overall score for breathlessness severity that incorporates seven physical items and five affective items
Pittsburgh sleep quality index | 6 weeks
  Pittsburgh sleep quality index (PSQI) is an effective instrument used to measure the quality and pattern of sleep. The PSQI was originally designed for use in clinical populations as a simple and valid assessment of both sleep quality and disturbance that might affect sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Ameena Amjad, tDPT, Principal Investigator — Riphah International University
Locations (1):
- Laeeque Rafiq Hospital, Lar, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toskala E, Kennedy DW. Asthma risk factors. Int Forum Allergy Rhinol. 2015 Sep;5 Suppl 1(Suppl 1):S11-6. doi: 10.1002/alr.21557. PMID 26335830
- [Background] Janson C, Accordini S, Cazzoletti L, Cerveri I, Chanoine S, Corsico A, Ferreira DS, Garcia-Aymerich J, Gislason D, Nielsen R, Johannessen A, Jogi R, Malinovschi A, Martinez-Moratalla Rovira J, Marcon A, Pin I, Quint J, Siroux V, Almar E, Bellisario V, Franklin KA, Gullon JA, Holm M, Heinrich J, Nowak D, Sanchez-Ramos JL, Weyler JJ, Jarvis D. Pharmacological treatment of asthma in a cohort of adults during a 20-year period: results from the European Community Respiratory Health Survey I, II and III. ERJ Open Res. 2019 Feb 1;5(1):00073-2018. doi: 10.1183/23120541.00073-2018. eCollection 2019 Feb. PMID 30723731
- [Background] Bruurs ML, van der Giessen LJ, Moed H. The effectiveness of physiotherapy in patients with asthma: a systematic review of the literature. Respir Med. 2013 Apr;107(4):483-94. doi: 10.1016/j.rmed.2012.12.017. Epub 2013 Jan 18. PMID 23333065
- [Background] Akgun Sahin Z, Dayapoglu N. Effect of progressive relaxation exercises on fatigue and sleep quality in patients with chronic obstructive lung disease (COPD). Complement Ther Clin Pract. 2015 Nov;21(4):277-81. doi: 10.1016/j.ctcp.2015.10.002. Epub 2015 Oct 19. PMID 26573455
- [Background] Santino TA, Chaves GS, Freitas DA, Fregonezi GA, Mendonca KM. Breathing exercises for adults with asthma. Cochrane Database Syst Rev. 2020 Mar 25;3(3):CD001277. doi: 10.1002/14651858.CD001277.pub4. PMID 32212422
- [Background] Pourdowlat G, Hejrati R, Lookzadeh S. The effectiveness of relaxation training in the quality of life and anxiety of patients with asthma. Adv Respir Med. 2019;87(3):146-151. doi: 10.5603/ARM.2019.0024. PMID 31282555
- [Background] Climaco DCS, Lustosa TC, Silva MVFP, Lins-Filho OL, Rodrigues VK, Oliveira-Neto LAP, Feitosa ADM, Queiroga FJP Jr, Cabral MM, Pedrosa RP. Sleep quality in COPD patients: correlation with disease severity and health status. J Bras Pneumol. 2022 Apr 29;48(3):e20210340. doi: 10.36416/1806-3756/e20210340. eCollection 2022. PMID 35508063
- [Background] Ebadi Z, Goertz YMJ, Van Herck M, Janssen DJA, Spruit MA, Burtin C, Thong MSY, Muris J, Otker J, Looijmans M, Vlasblom C, Bastiaansen J, Prins J, Wouters EFM, Vercoulen JH, Peters JB. The prevalence and related factors of fatigue in patients with COPD: a systematic review. Eur Respir Rev. 2021 Apr 13;30(160):200298. doi: 10.1183/16000617.0298-2020. Print 2021 Jun 30. PMID 33853886
- [Background] James MD, Milne KM, Phillips DB, Neder JA, O'Donnell DE. Dyspnea and Exercise Limitation in Mild COPD: The Value of CPET. Front Med (Lausanne). 2020 Aug 13;7:442. doi: 10.3389/fmed.2020.00442. eCollection 2020. PMID 32903547
- [Background] Lu Y, Li P, Li N, Wang Z, Li J, Liu X, Wu W. Effects of Home-Based Breathing Exercises in Subjects With COPD. Respir Care. 2020 Mar;65(3):377-387. doi: 10.4187/respcare.07121. Epub 2019 Nov 12. PMID 31719191
- [Background] Setyowati A, Chung MH. Validity and reliability of the Indonesian version of the Pittsburgh Sleep Quality Index in adolescents. Int J Nurs Pract. 2021 Oct;27(5):e12856. doi: 10.1111/ijn.12856. Epub 2020 Jul 7. PMID 32632973
- [Background] Shi C, Goodall M, Dumville J, Hill J, Norman G, Hamer O, Clegg A, Watkins CL, Georgiou G, Hodkinson A, Lightbody CE, Dark P, Cullum N. The accuracy of pulse oximetry in measuring oxygen saturation by levels of skin pigmentation: a systematic review and meta-analysis. BMC Med. 2022 Aug 16;20(1):267. doi: 10.1186/s12916-022-02452-8. PMID 35971142
- [Background] Yorke J, Swigris J, Russell AM, Moosavi SH, Ng Man Kwong G, Longshaw M, Jones PW. Dyspnea-12 is a valid and reliable measure of breathlessness in patients with interstitial lung disease. Chest. 2011 Jan;139(1):159-64. doi: 10.1378/chest.10-0693. Epub 2010 Jul 1. PMID 20595454
- [Background] Holloway EA, West RJ. Integrated breathing and relaxation training (the Papworth method) for adults with asthma in primary care: a randomised controlled trial. Thorax. 2007 Dec;62(12):1039-42. doi: 10.1136/thx.2006.076430. Epub 2007 Jun 15. PMID 17573445